CLINICAL TRIAL: NCT05326633
Title: Effect of Protein, Mobility Therapy and Electric Stimulation on Recovery in Older Survivors of Critical Illness
Brief Title: Effect of Protein, Mobility Therapy and Electric Stimulation on Recovery in Older ICU Survivors
Acronym: ProMoTE
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Avelino Verceles, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00083098
Record Dates: First submitted 2022-02-07; First posted 2022-04-13 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Critical Illness; Sarcopenia; ICU Acquired Weakness
Keywords: ICU Acquired Weakness; Critical Care; Long Term Acute Care Hospital; Protein; Neuromuscular electric stimulation; Physical Rehabilitation; Geriatric population
MeSH Terms: conditions — Critical Illness; Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- UC only (No Intervention): LTACH control group receiving usual care (UC) only.
- MRP+HPRO+NMES+UC (Active Comparator): LTACH group receiving mobility based rehabilitation (MRP) + neuromuscular electric stimulation (NMES) + high protein supplementation (HPRO) + usual care (UC)
  Interventions: Combination Product: MRP and High Protein Supplement (HPRO) and Neuromuscular Electric Stimulation (NMES)

INTERVENTIONS:
Combination Product: MRP and High Protein Supplement (HPRO) and Neuromuscular Electric Stimulation (NMES) — Mobility-based physical rehabilitation sessions performed 5 times/week by a study PT to provide strength and cardiopulmonary endurance training. High whey protein shakes prescribed to a total intake of 1.6-1.8 g/kg/d in 2 divided doses based on caloric needs. 2 x 30-minute lower extremity electric stimulation sessions/day, 5 times/wk performed by study PT.
  Arms: MRP+HPRO+NMES+UC

SUMMARY:
Older ICU survivors with ICU acquired weakness (ICUAW) are malnourished, sarcopenic, and functionally debilitated as a consequence of the high burden of comorbidities common in the elderly. To address the sequalae of critical illnesses, the investigators will perform a trial incorporating an intervention that combines mobility-based physical rehabilitation (MRP), high protein supplementation (HPRO), and neuromuscular electric stimulation (NMES). The investigators will then assess both clinical and functional outcomes and determine the relationship of disability with systemic inflammation.

DETAILED DESCRIPTION:
Annually, nearly 3 million patients ≥ 65 years old are admitted to intensive care units (ICUs) nationwide, 20% of whom experience a long, protracted ICU stay resulting in muscle deconditioning, atrophy, inflammation, and functional disability necessitating transfer from the ICU to a long term acute care hospitals (LTACH). In the LTACH exacerbations of chronic comorbidities and the cycle of prolonged bed rest, ongoing inflammation and malnutrition often leads to continued functional disability, immobility, prolonged mechanical ventilation and increased one-year mortality of up to 25%. After a patient has survived critical illness and is transferred to an LTACH facility, one of the major challenges of their continued care is how to address - and ameliorate - their profound physical and functional deficits.

To address these sequalae of chronic critical illness, the investigators will perform a trial incorporating an intervention that combines mobility-based physical rehabilitation (MRP), high protein supplementation (HPRO) and neuromuscular electric stimulation (NMES) to assess both clinical and functional outcomes and to determine the relationship of disability with systemic inflammation. The investigators will prospectively randomize patient to receive our multicomponent intervention or usual care and assess the outcomes of functional mobility, change in muscle mass and discharge disposition. Additionally, the investigators will determine the effects of our intervention on inflammatory cytokine profiles to determine to what degree systemic inflammation mediates clinical recovery.

ELIGIBILITY:
Inclusion Criteria:

1. LTACH admission within 72 hours
2. Age ≥ 60 years old
3. Prior ICU stay ≥ 2 weeks
4. Able to follow commands in English
5. Pre-ICU Barthel Index ≥ 70
6. Able to give consent
7. Able to perform physical therapy
8. All four limbs intact and mobile prior to LTACH admission

Exclusion Criteria:

1. Acute kidney injury with a glomerular filtration rate <15 ml/min
2. Diagnosis of severe organ dysfunction including end stage liver disease or cirrhosis
3. Diagnosis of active cancer
4. Severe functional impairment or physical impairment to rehabilitation
5. Liver function tests >2.5x normal limits
6. Chronic dementia or cognitive impairment

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle mass | Days 0 to 14 to 28
  Muscle mass will be measured by lower extremity muscle CT scans to calculate muscle volume and cross sectional area.
Change in Muscle strength | Days 0, 7, 14, 21 and 28
  Handgrip strength obtained using a hand grip dynamometer and manual muscle testing using hand held dynamometer
Change in Systemic Inflammation | Days 0, 7, 14, 21 and 28
  Quantitative analysis of CRP, IFN-γ, IL-1α, IL-1β, IL-6, and IL-8.

SECONDARY OUTCOMES:
Change in Functional status - SPPB | Days 0, 7, 14, 21 and 28
  Functional status will be assessed by using the Short Physical Performance Battery (SPPB)
Change in Functional status - FSS-ICU | Days 0, 7, 14, 21 and 28
  Functional status will be assessed by using the Functional Status Score in the ICU (FSS-ICU).
Change in Mobility status - ICU mobility Scale | Days 0, 7, 14, 21 and 28
  Mobility status will be assessed weekly using the 1-item ICU Mobility Scale weekly in those physically capable.
Change in Mobility status - 6 minute walk distance | Days 0, 7, 14, 21 and 28
  Mobility status will be assessed weekly using the total 6 Minute Walk distance in those physically capable.
Change in Mobility status - gait speed | Days 0, 7, 14, 21 and 28
  Mobility status will be assessed weekly using gait speed in those physically capable.
Discharge disposition (LTACH to home, nursing home, acute rehabilitation, readmission, or death) | up to or after Day 28
  Discharge disposition from the LTACH to home, nursing home, acute rehabilitation, readmission, or death)

CONTACTS AND LOCATIONS:
Locations (1):
- U of Maryland, Baltimore, Professional Schools IRB, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No